CLINICAL TRIAL: NCT02352610
Title: A Prospective Randomized Trial Comparing Standard Ligament Reconstruction Tendon Interposition (LRTI) VS Ligament Reconstruction Tendon Interposition (LRTI) With an Interference Screw for Thumb Carpometacarpal Arthritis - Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Andrew Trenholm (Other)
Responsible Party: Sponsor-Investigator, Andrew Trenholm, Orthopaedic Surgeon, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-239
Record Dates: First submitted 2015-01-08; First posted 2015-02-02 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Osteoarthritis
Keywords: carpometacarpal joints
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LRTI without a Biotenodesis Screw (Active Comparator): Ligament Reconstruction Tendon Interposition without a Biotenodesis Screw
  Interventions: Procedure: LRTI
- LRTI with Biotenodesis Screw (Active Comparator): Ligament Reconstruction Tendon Interposition with Biotenodesis Screw
  Interventions: Procedure: LRTI; Device: Biotenodesis Screw

INTERVENTIONS:
Procedure: LRTI
Device: Biotenodesis Screw
  Arms: LRTI with Biotenodesis Screw

SUMMARY:
A Prospective Randomized Trial Comparing Standard Ligament Reconstruction Tendon Interposition (LRTI) VS Ligament Reconstruction Tendon Interposition (LRTI) with an interference screw for thumb carpometacarpal arthritis

DETAILED DESCRIPTION:
This study will be a prospective randomized trial done in a single academic center. The patients who meet the inclusion criteria and agree to participate in the trial will be scheduled for a first CMC joint procedure. The procedure, standard LRTI or LRTI with a biotenodesis screw, will be allocated in a randomized fashion in the operating room using a sealed opaque envelope. After the surgery the patient will be placed in a spica splint for 1-2 weeks. Following suture removal, a thumb spica cast will be applied for immobilization for a total of 6 weeks of post-operative immobilisation.

The potential population for this study will include all patients with first carpometacarpal joint arthritis that have failed a conservative treatment. The primary outcome will be the thumb subsidence measured as the percentage of trapezial height, which correlates with stability. Subsidence will be measured on stress x-ray under a standard pinch load. Secondary outcomes will be function measured in 4 different ways: the range of motion compared to the contralateral side, pinch and grip strength compared to the other side, the Disabilities of the Arm Shoulder and Hand (DASH) score and the pain score on a visual analogue scale.

ELIGIBILITY:
Inclusion Criteria:

* First CMC primary osteoarthritis refractory to conservative treatment
* Patient >age 18
* Able to read and understand English
* Available for 2 year follow up

Exclusion Criteria:

* Inflammatory Arthritis
* Active infection in the first CMC joint
* Concomitant neuropathy
* Previous surgical procedure on the thumb
* Active or status post CRPS
* Severe ¨Z ¨deformity that requires palmar plate advancement
* Unwilling to participate in a research project
* Contralateral first CMC joint surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-03; Primary Completion 2018-02-22 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Subsidence of CMC joint | 6 weeks, 3 months, 6 months, 1 year, 2 years
  Measurement of trapezial height as a percentage of pre-operative height

SECONDARY OUTCOMES:
EQ-5D Health Questionnaire Score | Baseline, 6 weeks, 3 months, 6 months, 1 year, 2 years
DASH questionnaire score | Baseline, 6 weeks, 3 months, 6 months, 1 year, 2 years
Grip strength as measured by dynamometer | Baseline, 3 months, 6 months, 1 year, 2 years
Pinch strength as measured by dynamometer | Baseline, 3 months, 6 months, 1 year, 2 years
Opposition as measured by goniometer | Baseline, 3 months, 6 months, 1 year, 2 years
  thumb range of motion
Radial abduction as measured by goniometer | Baseline, 3 months, 6 months, 1 year, 2 years
  thumb range of motion
Palmar abduction as measured by goniometer | Baseline, 3 months, 6 months, 1 year, 2 years
  thumb range of motion
Pain score on the visual analogue scale | Baseline, 2 weeks, 6 weeks, 3 months, 6 months, 1 year, 2 years
  visual analogue scale

OTHER OUTCOMES:
Number of participants with Adverse Events | Baseline, 2 weeks, 6 weeks, 3 months, 6 months, 1 year, 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia, Canada